CLINICAL TRIAL: NCT01306994
Title: Freeman-Sheldon Syndrome Evaluation and Diagnosis in Clinical Settings (FSS-EDICT) I: a Case-Control, Cross-Sectional Study of Baseline and Stress Physiology Parameters
Brief Title: Study of Resting and Exercising Body Functioning in Freeman-Sheldon Syndrome and Related Conditions
Acronym: FSS-EDICT I
Status: Withdrawn | Type: Observational
Why Stopped: Lack of patient interest
Sponsor: Freeman-Sheldon Research Group, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 000079; U1111-1120-5931 (Other: World Health Organisation, Universal Trial Number)
Record Dates: First submitted 2011-02-26; First posted 2011-03-02 (Estimated); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Arthrogryposis; Craniofacial Abnormalities
Keywords: Exercise Test; Bicycle Ergometry Test; Stress Test
MeSH Terms: conditions — Arthrogryposis; Craniofacial Abnormalities | interventions — Lactic Acid; Glucose; Hematologic Tests; Adenosine Triphosphate; Glucose Tolerance Test; Blood Glucose; Exercise Test; Health Records, Personal; Restraint, Physical; Independent Medical Evaluation; Gait Analysis; Interview, Psychological

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Blood samples will be taken but no retention is expected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Syndrome Group: Individuals with Freeman-Sheldon, Sheldon-Hall, distal arthrogryposis type 1, or distal arthrogryposis type 3
  Interventions: Other: Lactate, Glucose, and Adenosine Triphosphate Blood Levels; Procedure: Physiological Stress Test; Other: Functional Enquiry Form; Other: Strength, Joint ROM, Girth and Length Measurements; Other: Study Physical Examination; Other: Observational Gait Analysis; Other: Mental Health Interview
- Control Group: Healthy individuals
  Interventions: Other: Lactate, Glucose, and Adenosine Triphosphate Blood Levels; Procedure: Physiological Stress Test; Other: Functional Enquiry Form; Other: Strength, Joint ROM, Girth and Length Measurements; Other: Study Physical Examination; Other: Observational Gait Analysis; Other: Mental Health Interview

INTERVENTIONS:
Other: Lactate, Glucose, and Adenosine Triphosphate Blood Levels — Completed during the clinical examination and exercise test by the researchers, lactate, glucose, and free and total adenosine triphosphate blood levels are determined at rest and during exercise.
  Other Names: ATP levels; ATP blood levels; adenosine triphosphate test; blood test for ATP; blood test for adenosine triphosphate; ATP blood test; adenosine triphosphate blood test; ATP test; glucose test; glucose blood test; sugar test; lactic acid levels; lactic acid blood test; lactate blood test; lactate levels
Procedure: Physiological Stress Test — During exercise, heart and lung function are monitored for changes caused by exercise, which increases the body's need for oxygen and puts extra demands on the heart. In this study, testing is done using a cycle ergometer and conducted according to the standardised exponential exercise protocol (STEEP).
  Other Names: stress test; graded exercise test; maximal exercise test; VO2 max test; maximal oxygen uptake test; exercise tolerance test; exercise stress test
Other: Functional Enquiry Form — Evaluated before clinical examination, it is a checklist of medical problems.
  Other Names: FSRG Form 08; health history; review of systems; systems review; medical history; personal health history
Other: Strength, Joint ROM, Girth and Length Measurements — Completed during the clinical examination by the researchers, it is a structured approach to evaluation of muscles, joints, arms, thighs, and legs.
  Other Names: SF 527; Standard Form 527; musculoskeletal examination; musculoskeletal exam; musculoskeletal evaluation; musculoskeletal assessment; extremity examination; extremity evaluation; extremity assessment; extremity exam
Other: Study Physical Examination — Completed during the clinical examination by the researchers, it is a structured approach to a full physical examination (minus breasts, genitalia, or rectum).
  Other Names: FSRG Form 14; physical examination; physical evaluation; physical assessment; medical examination; medical evaluation; medical assessment; full medical examination; full medical evaluation; full medical assessment; periodic medical examination; periodic medical evaluation; periodic medical assessment; annual medical examination; annual medical evaluation; annual medical assessment; yearly medical examination; yearly medical evaluation; yearly medical assessment; full physical examination; full physical evaluation; full physical assessment; complete physical examination; complete physical evaluation; complete physical assessment; yearly physical examination; yearly physical evaluation; yearly physical assessment; annual physical examination; annual physical evaluation; annual physical assessment; periodic physical examination; periodic physical evaluation; periodic physical assessment; screening physical examination; screening physical evaluation; screening physical assessment; screening physical; physical; periodic physical; annual physical; annual check-up; annual check up; yearly physical; yearly check up; yearly check-up; check up; check-up; medical check-up; medical check up; annual medical check-up; annual medical check up; yearly medical check-up; yearly medical check up; periodic medical check-up; periodic medical check up; periodic health evaluation; periodic health assessment; annual health evaluation; annual health assessment; yearly health evaluation; yearly health assessment; screening health evaluation; screening health assessment; screening medical examination; screening medical evaluation; screening medical assessment; med check
Other: Observational Gait Analysis — Completed during the clinical examination by researchers, it is a structured approach to evaluation of a person's walking.
  Other Names: FSRG 10; gait analysis; functional gait analysis
Other: Mental Health Interview — Completed during the clinical examination by the researchers, it is a general evaluation of mental health status.
  Other Names: psychiatric examination; psychiatric evaluation; psychiatric assessment; psychiatric interview; diagnostic mental health examination; diagnostic mental health evaluation; diagnostic mental health assessment; diagnostic psychiatric examination; diagnostic psychiatric evaluation; diagnostic psychiatric assessment; diagnostic psychiatric interview; intake examination; intake evaluation; intake assessment; intake interview; mental health evaluation; mental health examination; mental health assessment; psychological examination; psychological evaluation; psychological assessment; psychological interview; psychological intake examination; psychological intake evaluation; psychological intake assessment; psychological intake interview

SUMMARY:
The hypotheses of the present study of Freeman-Sheldon syndrome (FSS) and related conditions are: (1) that exercise capacity is lower in FSS patients versus normal controls, and the lower exercise capacity is due to changes in the muscles' normal structure and an inability of sufficient quantity of the energy molecule to bind to muscle; (2) this muscle problem reduces amount of air that can get in the lung and amount of oxygen carried in the blood, which then has the effect of increasing heart and respiration rates, blood pressure, and deep body temperature, and produces muscle rigidity; (3) the events noted above, when they occur during cardiac stress testing, are related to a problem similar to malignant hyperthermia (MH) reported in some muscle disorders without use of drugs known to cause MH. MH (a life-threatening metabolic reaction that classically is triggered when susceptible persons receive certain drugs used in anaesthesia.

DETAILED DESCRIPTION:
This study is a research project initiated by the graduate research student (Mikaela I. Poling) and assisted by the clinical genetics fellow and graduate student (Andrés Morales) in partial fulfilment the requirements for their Masters degrees in Clinical and Applied Physiology, under approval, direction, and supervision of the study PI (Rodger J. McCormick).

Importance of Present Study:

FSS is a rare human neuromusculoskeletal disorder present before birth, involving primarily limb and craniofacial deformities. There are no prospective studies addressing physiological parameters, which are necessary to enable understanding of the underlying pathology and pathophysiology of Freeman-Sheldon syndrome. Elucidating any deviations in baseline and stress physiological parameters in FSS patients versus standard normal values and normal control subjects is of critical importance in tailoring therapeutic interventions to this challenging patient population.

Background:

Vanek et al. (1986) purposed FSS spectrum is a non-progressive congenital myopathy, giving pathological and electromyographical (EMG) evidence. They found white fibrose tissue within histologically normal muscle fibres, resulting in abnormal EMGs.

Toydemir et al. (2006) showed that mutations in embryonic myosin heavy chain 3 (MYH3), caused classic FSS phenotype, in which they screened 28 probands. In 20 patients, new missense mutations caused substitution of arginine at position 672 (arg672) by histidine or cytosine; arg672 is found in all myosin proteins post-embryonically. Of the remaining six patients in whom mutations were found, three had new missense or familial mutations; three other patients with sporadic expression had new, which were also found in Sheldon-Hall syndrome (SHS); two patients had no recognized mutations. They postulated these allelic variations at arg672 could affect adenosine triphosphate (ATP) binding. It is unknown how these mutations might correlate to the phenotypes observed. Their laboratory, including Stevenson et al. (2006) also presented strong evidence that FSS and SHS and similar distal arthrogryposes (DA) were distinct entities based on phenotype, natural history, and genotype.

Portillo et al. (unpublished data), in study of biopsies from their patient, found no evidence of muscle in the superior orbicularis oculi and found highly variable fibre size as a single pathological feature in a single vastus lateralis biopsy. Clinically, their patient, who had to-date the most severe expression of FSS, exhibited no function of the superior eyelid and reasonable muscle tone, bulk, and strength in the thigh. These findings suggested variable syndromic affectation by body region. They reported exertional dyspnea and resting tachycardia, without pathological features, in their patient and anecdotal information concerning exertional dyspnea in two other adult FSS patients. They also documented the occurrence of unexplained, seemingly stress-induced, episodic fever in their patient that resembled the malignant hyperthermia (MH) clinical triad of hyperthermia, tachycardia, and muscle rigidity.

In addition to age, gender, physical activity status, and concomitant disease and disability, maximal oxygen uptake, a function of exercise capacity, is genetically-controlled, and as already documented in other muscle disorders, the idiopathic febrile episodes reported by Portillo et al. may share physiological and biochemical similarities to the well-defined congenital muscle anomaly MH, which classically occurs when susceptible individuals receive inhaled anaesthetics, such as ether and halothane, or depolarizing muscle relaxants during surgery. Together, these clinical observations suggested there may be some syndromic relationship to exercise capacity and development of MH-like febrile syndrome, and it will be important to demonstrate these findings in a controlled experimental setting.

Significant differences among the similar distal arthrogryposes (DAs) may exist, with respect to the above, and this will be important to define experimentally, as well. Data concerning baseline and stress physiology in FSS and similar DAs could help to further define the distinct DA phenotypes clinically similar to FSS, contributing to nosological classification of FSS and related entities. This study will include FSS, Sheldon-Hall syndrome, DA type 1, and DA type 3.

ELIGIBILITY:
Syndrome Group Inclusion Criteria:

* Freeman-Sheldon syndrome,
* Sheldon-Hall syndrome,
* Distal arthrogryposis type 1, or
* Distal arthrogryposis type 3
* Deceased patients with enough clinical information available to satisfy study requirements

Syndrome Group Exclusion Criteria:

* Individuals not confirmed to have a condition under study
* Deceased patients without enough clinical information available to satisfy study requirements
* Patients with other anomalies, not having one of the above syndromes
* Patients or parents of minor children not willing to give consent
* Mature female patients who are pregnant or breast-feeding will be reassessed for consideration for enrolment.
* Mature female patients who are currently experiencing menses will be reassessed for consideration for enrolment.
* Patients with active, acute comorbid illness will be reassessed for consideration for enrolment.

Control Group Inclusion Criteria:

* Subjects must be healthy and free of active disease.
* Subject or parent of minor child must be willing to give consent.
* Subjects must fall within the age-bracket to be matched with a Syndrome Group patient already screened and enroled in the study
* Subjects must be non-tobacco users and non-drinkers.

Control Group Exclusion Criteria:

* Subjects exceptional for their age in body weight, stature, or habitus according to commonly accepted guidelines
* Subjects with active psychiatric illness, as manifested by abnormal mental status examination
* Subjects with active physical illness, especially respiratory or cardiac problem, as manifested by abnormal findings on physical examination
* Subjects with significant diagnosis of a constitutional disease or genetic disorder
* Subjects with a history of severe trauma resulting in either an anatomical of physiological deformity that impairs function
* Non-living subjects
* Candidates who fail the stress test
* Mature female subjects who are pregnant or breast-feeding will be reassessed for consideration for enrolment.
* Mature female subjects who are currently experiencing menses will be reassessed for consideration for enrolment.
* Subjects with active, acute illness will be reassessed for consideration for enrolment.
* Any other condition or anomaly expected to affect current physiology listed in AFI-48-123.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients world-wide are welcome, so-long as they have a qualifying diagnosis. Healthy controls are welcome world-wide, as well.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Heart rate | Evaluated at rest and while exercising, during two study visits (lasting an average of 1-3 hours)
  Increased heart rate, measured electrocardiographically, is used as an index of cardiovascular strain imposed by needs during exercise and exaggerated by Freeman-Sheldon and related conditions.
Oxygen Consumption | Evaluated at rest and while exercising, during two study visits (lasting an average of 1-3 hours)
  Oxygen consumption, measured by ventilation of expired oxygen, is used as a measure of physiological strain imposed by metabolic needs during exercise and exaggerated by Freeman-Sheldon and related conditions.

SECONDARY OUTCOMES:
Non-Invasive Arterial Blood Pressure | Evaluated at rest and while exercising, during two study visits (lasting an average of 1-3 hours)
  Increased non-invasive arterial blood pressure rate is used as an index of cardiovascular strain imposed by needs during exercise and exaggerated by Freeman-Sheldon and related conditions.
Spirometry (Forced Expiratory Volume/Forced Vital Capacity) | Evaluated before and after exercise, during two study visits (lasting an average of 1-3 hours)
  Decreased ability of the lungs to move air, measured by forced expiration, is used as an index of strain imposed by Freeman-Sheldon syndrome and related conditions.
Saturation of Peripheral Oxygen | Evaluated at rest and while exercising, during two study visits (lasting an average of 1-3 hours)
  Decreased saturation of peripheral oxygen, measured by pulse oxymetry, is used as a measure of physiological strain imposed by metabolic needs during exercise and exaggerated by Freeman-Sheldon and related conditions.
Respiratory Rate | Evaluated at rest and while exercising, during two study visits (lasting an average of 1-3 hours)
  Increased respiratory rate, measured by plethysmograph, is used as a measure of physiological strain imposed by metabolic needs during exercise and exaggerated by Freeman-Sheldon and related conditions.
Heart Rhythm | Evaluated at rest and while exercising, during two study visits (lasting an average of 1-3 hours)
  Heart rhythms, monitored by electrocardiograph, are used as an index of cardiovascular strain imposed by needs during exercise and exaggerated by Freeman-Sheldon and related conditions.
Core Temperature | Evaluated at rest and while exercising, during two study visits (lasting an average of 1-3 hours)
  Increased core temperature, measured as oesophageal temperature, is used as a measure of physiological strain imposed by metabolic needs during exercise and exaggerated by Freeman-Sheldon, related conditions, and malignant hyperthermia.
Adenosine Triphosphate | Evaluated at rest and while exercising, during two study visits (lasting an average of 1-3 hours)
  Decreased adenosine triphosphate, measured as capillary blood level, is used as a measure of physiological strain imposed by metabolic needs during exercise and exaggerated by Freeman-Sheldon and related conditions.
Perceived Exertion | Evaluated at rest and while exercising, during two study visits (lasting an average of 1-3 hours)
  Increased perceived exertion, measured using the Borg scale, are used as an index of fatigue.
Muscle Rigidity | Evaluated while exercising, during second of two study visits (lasting an average of 1-3 hours)
  Increased muscle rigidity, evaluated by clinical examination and patient self-report, is used as an indicator of malignant hyperthermia, when increased core temperature, heart rate, and respiratory rate are present.
Functional and Health-Related Quality of Life | Evaluated in first of two study visits, lasting an average of 1-3 hours
  Functional and health-related quality of life, measured with the Medical Outcomes Trust Short Form (36) Health Survey (SF-36), is used as a general prediction of expected physical exercise capacity.
Lactic Acid | Evaluated at rest and while exercising, during two study visits (lasting an average of 1-3 hours)
  Lactic acid, measured by capillary blood level, is used as a measure of physiological strain imposed by metabolic needs during exercise and exaggerated by Freeman-Sheldon and related conditions.
Glucose | Evaluated at rest and while exercising, during two study visits (lasting an average of 1-3 hours)
  Glucose, measured by capillary blood level, is used as an index of physiological strain, together with lactic acid and adenosine triphosphate capillary blood levels, imposed by metabolic needs during exercise and exaggerated by Freeman-Sheldon and related conditions.

OTHER OUTCOMES:
Body Composition | Evaluated before exercise, during two study visits (lasting an average of 1-3 hours)
  Body composition, measured by calliper, together with direct indices of physiological strain, is used to determined metabolic disease burden of Freeman-Sheldon syndrome and related conditions.
Hand Grip Strength | Evaluated during the first of two study visits
  Decreased hand grip strength, measured by a hand dynamometer, is used as an index of physiological strain imposed by Freeman-Sheldon and related conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Freeman-Sheldon Research Group, Inc. Headquarters, Buckhannon, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No
We do not intend to share any individual participant data.

REFERENCES:
- [Background] Vanek J, Janda J, Amblerova V, Losan F. Freeman-Sheldon syndrome: a disorder of congenital myopathic origin? J Med Genet. 1986 Jun;23(3):231-6. doi: 10.1136/jmg.23.3.231. PMID 3723551
- [Background] Toydemir RM, Rutherford A, Whitby FG, Jorde LB, Carey JC, Bamshad MJ. Mutations in embryonic myosin heavy chain (MYH3) cause Freeman-Sheldon syndrome and Sheldon-Hall syndrome. Nat Genet. 2006 May;38(5):561-5. doi: 10.1038/ng1775. Epub 2006 Apr 16. PMID 16642020
- [Background] Stevenson DA, Carey JC, Palumbos J, Rutherford A, Dolcourt J, Bamshad MJ. Clinical characteristics and natural history of Freeman-Sheldon syndrome. Pediatrics. 2006 Mar;117(3):754-62. doi: 10.1542/peds.2005-1219. PMID 16510655
- [Background] Portillo AL, Chamberlain RL, McCormick RJ, Poling MI. Histopathological and Operative Findings in a Severe Case of Freeman-Sheldon Syndrome: Implications for Nosology and Therapy. (Unpubl.) 2010.
- [Background] Litman RS, Rosenberg H. Malignant hyperthermia: update on susceptibility testing. JAMA. 2005 Jun 15;293(23):2918-24. doi: 10.1001/jama.293.23.2918. PMID 15956637
- [Background] McCormick RJ. A Proposal for a Thesis: Heat Tolerance in Exercising Lean and Obese Middle-Aged Men. DEd diss., the Pennsylvania State University, 1973.
- [Background] Myhill S, Booth NE, McLaren-Howard J. Chronic fatigue syndrome and mitochondrial dysfunction. Int J Clin Exp Med. 2009;2(1):1-16. Epub 2009 Jan 15. PMID 19436827
- [Background] Northridge DB, Grant S, Ford I, Christie J, McLenachan J, Connelly D, McMurray J, Ray S, Henderson E, Dargie HJ. Novel exercise protocol suitable for use on a treadmill or a bicycle ergometer. Br Heart J. 1990 Nov;64(5):313-6. doi: 10.1136/hrt.64.5.313. PMID 2245110
- [Background] Franklin B, Fern A, Fowler A, Spring T, Dejong A. Exercise physiologist's role in clinical practice. Br J Sports Med. 2009 Feb;43(2):93-8. doi: 10.1136/bjsm.2008.055202. Epub 2008 Dec 2. PMID 19050005